CLINICAL TRIAL: NCT00959010
Title: Biochemical Effects of a Long-term Supplementation With Omega-3 Polyunsaturated Fatty Acids in Cystic Fibrosis
Brief Title: Omega 3 Supplementation in Cystic Fibrosis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Queen Fabiola Children's University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HU01/PNE/MUCO1; 2006-004155-38
Record Dates: First submitted 2009-08-13; First posted 2009-08-14 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Cystic Fibrosis
Keywords: Omega 3; Cystic Fibrosis; Inflammatory markers
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Omega 3 Premium (Experimental): capsules containing 300mg of omega-3 triglycerides with 100mg DHA and 150mg EPA
  Interventions: Dietary Supplement: omega-3 triglycerides
- Placebo (Placebo Comparator): capsules containing middle chain triglycerides
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: omega-3 triglycerides — capsules containing 300mg of omega-3 triglycerides with 100mg DHA and 150mg EPA, 60mg/kg/day 3 times a day during 12 months.
  Arms: Omega 3 Premium
Dietary Supplement: Placebo — capsules containing middle chain triglycerides
  Arms: Placebo

SUMMARY:
Essential fatty acids (EFA) deficiency has been often reported in patients with cystic fibrosis (CF), particularly in those homozygous for the DF508 mutation. Clinical symptoms of CF may be influenced by correcting EFA deficiency. Nevertheless, the value of EFA supplementation in CF remains controversial. Within this multicentric and international randomized placebo-controlled trial it will be evaluated, according to recommendations of Cochrane analysis, beneficial effects of an oral supplementation with polyunsaturated fatty acids on selected biochemical and functional outcome parameters such as inflammatory biomarkers, incorporation into cell membrane phospholipids, lung function, exercise tolerance, clinical and nutritional status and properties of transepithelial ion transport. The study will be undertaken in a cohort of CF patients aged over 6 years old (60 patients), homozygous for the DF508 mutation and treated by Azithromycine. Supplementation will be performed with a triglyceride source at a daily dose of 60 mg/kg of omega-3 polyunsaturated fatty acids (Omega 3 Premiumâ, Laboratoires Ponroy, France). Before enrolled into the trial and during the study, patients will undergo nutritional assessment by evaluation of total and fat dietary intake and overall calorie intake using a 3-days diet records and a food frequency questionnaire. Plasma and erythrocyte membrane EFA profiles and inflammatory markers will be monitored in baseline conditions, at 3, at 6 and 12 months after starting the treatment. Lung function will be performed at each patient visit and an exercise test will be done before and at the end of the treatment. Properties of ion transport will be searched by sweat testing before and at the end of the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient over 6 years of age at visit 1 with stable cystic fibrosis
2. Documented Homozygous for DeltaF508 mutation
3. Patient treated with stable dose of Azithromycine since at least 3 months
4. Able to perform pulmonary function test and swallow capsules
5. Female patient of childbearing potential must have a negative serum pregnancy test prior to enrolment and must agree to practice effective birth control during the study and 6 weeks thereafter
6. Signed informed consent obtained from the patient, or in case the patient is minor,from patient's legally acceptable representative (parents or guardians) according to ICH & local regulations. Child assent will be nevertheless obtained

Exclusion Criteria:

1. Ongoing acute illness including acute upper or lower respiratory infections within 2 weeks before baseline evaluation.
2. Abnormalities on screening chest x-ray (or CT-scan) suggesting clinically active pulmonary disease other than CF, or new, significant abnormalities such as atelectasis or pleural effusion which may be indicative of clinically active pulmonary involvement secondary to CF.
3. Any chronic (> 1 week daily) oral or intravenous inflammatory treatment, other than Azithromycine, given to the patient within 3 months before start of study treatment.
4. Active bleeding or increased risk of bleeding (rate of platelets < 50,000/mm3,patient treatment by anticoagulant or antiplatelet agents, disturbances of haemostasis with PTT <70%, bleeding disorders).
5. Patient has significant liver disease, defined as having elevated liver function tests with values 2-fold higher than the upper normal range of the investigational local lab or having abnormal ultrasound such as signs of cirrhosis.
6. Hypercholesterolemia (>240mg%).
7. Patient is pregnant or a breast-feeding mother
8. Patient is participating or has participated in another investigational drug trial or is receiving or has received an investigational drug within the last 28 days before entry into this study.
9. Patient is unlikely to comply with the visits scheduled in the protocol or enable to follow the study procedure.

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2008-10; Primary Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
LTB4/LTB5 ratio from baseline to the end of treatment assessment. | Assessment at 3-6-12 months

SECONDARY OUTCOMES:
To explore the change in other inflammatory biomarkers such as TNF-alpha, IL-6, IL-8, IL-17 & alpha-1 anti-trypsin. | Assessments at 3-6 and 12 months
To evaluate the incorporation into cell membrane phospholipids. | Assessments at 3-6-12 months
To evaluate the effects on the pulmonary function (FEV1) and on the exercise tolerance (VO2 max). | Assessment at 12 months
To evaluate the effects on the clinical status and the nutritional status. | Assessments at 3-6-9 and 12 months
To investigate the properties of transepithelial ion transport (sweat test). | Assessments at 12 months
To evaluate the long term overall safety and tolerability of Omega-3 EFA supplementation in CF patients. | Assessment at 3-6-9 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Hanssens, MD, Principal Investigator — Queen Fabiola Children's University Hospital
Locations (1):
- Hôpital Universitaire Des Enfants Reine Fabiola, Brussels, Belgium